CLINICAL TRIAL: NCT04713488
Title: An Open Study on the Safety, Tolerability, and Immunogenicity of "Sputnik Light" t Vaccine for Prevention of Coronavirus Infection Caused by the SARS-CoV-2 Viruso
Brief Title: An Open Study on the Safety, Tolerability, and Immunogenicity of "Sputnik Light" Vaccine
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Gamaleya Research Institute of Epidemiology and Microbiology, Health Ministry of the Russian Federation (Other)
Collaborators: Russian Direct Investment Fund (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 06 - Sputnik Light - 2020
Record Dates: First submitted 2021-01-13; First posted 2021-01-19 (Actual); Last update posted 2021-02-02 (Actual); Status verified 2021-01

CONDITIONS: COVID-19 Prevention
Keywords: COVID-19; vaccine; vector vaccine; Immunologic Factors; SARS-CoV-2
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sputnik Light Vaccine (Experimental): solution for intramuscular injection Composition for 1 dose (0.5 ml): Active substance: recombinant serotype 26 adenoviral particles containing the SARS-CoV-2 S protein gene, in the amount of (1.0±0.5) x 10*11 particles per dose.
  Interventions: Biological: Sputnik Light

INTERVENTIONS:
Biological: Sputnik Light — solution for intramuscular injection Composition for 1 dose (0.5 ml)
  Other Names: vector vaccine to help prevent the SARS-CoV-2-induced coronavirus infection

SUMMARY:
Phase I-II open prospective, two-stage, non-randomized study in healthy volunteers.

DETAILED DESCRIPTION:
Screening Period = up to 7 days All screening procedures must be executed within the shortest possible time frame before the scheduled date for Visit 1 (drug administration). The laboratory and instrumental examination data obtained within 14 days before the screening will be recorded as the screening data.

The trial will include 110 volunteers that will be administered the study drug. Outpatient observation will be done over the course of 4 visits: on day 10, 28, and 42 following drug administration Along with that, the study will be continued in accordance with the Protocol, accompanied by all the prescribed procedures and visits up to 180 days of observation.

Visit No. 0 (outpatient): screening Visit No. 1 (outpatient): vaccination Visits No. 2, 3, 4, 5, and 8: follow-up on days 10, 28, 42, 90, and180 after vaccination.

On days 120 and 150, visits 6 and 7 will be accomplished by telephone contact / telemedicine conference or, if necessary, in the form of an in-person visit.

Any volunteer who received a dose of the study drug will be registered as a trial participant, and his/her data will be used to help assess the drug's safety and tolerability.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent given by the subject to participate in the trial;
2. Males and females aged 18 years old and older
3. Lack of COVID-2019 in medical history: negative IgM and IgG SARS CoV2 antibodies enzyme-linked immunosorbent assay test result (no more than 14 days before being included in the trial)
4. Negative COVID-2019 PCR test result during the screening visit
5. No contact with COVID-2019-infected persons within at least 14 days before being included in the trial (according to what trial subjects state);
6. Negative HIV and hepatitis test results;
7. Consent to use effective contraception methods during the trial
8. Negative drugs or psychostimulants urine test during the screening visit;
9. Negative alcohol test during the screening visit;
10. Negative test for pregnancy (done for women with preserved reproductive potential)
11. No evident vaccine-induced reactions or complications after receiving immunobiological products in the person's medical history;
12. No acute infectious and/or respiratory diseases within at least 14 days before being included in the trial

Exclusion Criteria:

1. Any vaccination / immunization performed within 14 days prior to enrollment in the study, or a planned vaccination within 14 days after being administered the study drug;
2. Steroid therapy (except hormonal contraceptives or drugs used as hormone replacement therapy for menopause) that has not been completed 30 days before enrollment;
3. Therapy with immunoglobulins or other blood products not completed 30 days before enrollment in the trial
4. Immunosuppressor therapy that was completed within 3 months before being included in the trial
5. A vaccination against COVID-2019 using any other drugs, including in the course of other clinical studies
6. Female subjects during pregnancy or breastfeeding (for women with preserved reproductive potential);
7. Acute coronary syndrome or stroke suffered less than one year before enrolling in the trial
8. Tuberculosis, chronic systemic infections;
9. Complicated allergic history (severe life-threatening allergic reactions), hypersensitivity or allergic reactions to the introduction of immunobiological drugs, known allergic reactions to the components of the drug, exacerbation of allergic diseases on the day of enrolling in the trial;
10. Neoplasms in a person's medical history (ICD codes C00-D09);
11. Donated blood or plasma (450+ ml) within 2 months before enrollment;
12. Splenectomy in the person's medical history;
13. Neutropenia (absolute neutrophil count <1,000 mm3), agranulocytosis, significant blood loss, severe anemia (hemoglobin <80 g/L), immunodeficiency in the medical history within 6 months before the enrollment;
14. Active form of a disease caused by the human immunodeficiency virus, syphilis, hepatitis B or C;
15. Anorexia, protein deficiency of any origin;
16. Large tattoos at the injection site (deltoid muscle area), which does not allow assessing the localized response to administering the study drug/placebo
17. Alcohol or drug addiction in the person's medical history;
18. Registered with a psychiatrist
19. Participation in any other interventional clinical Trial within 90 days before the start of this trial
20. Any other condition that the researching physician considers to be a hindrance to completing the trial as per the protocol;
21. Research facility staff and other employees directly involved in the trial (research team members) and their families.
22. Any related conditions that, in the opinion of the study physician, could serve as a hindrance to participating in the trial.

Ages: 18 Years to 111 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2021-01-15 (Actual); Primary Completion 2021-07-20 (Estimated); Study Completion 2021-07-31 (Estimated)

PRIMARY OUTCOMES:
Changing of antibody levels against the SARS-CoV-2 glycoprotein S | at days 0,10, 28, 42, 180
  Determination of antibody levels against the SARS-CoV-2 glycoprotein S measured by an ELISA vs. baseline values
Number of Participants With Adverse Events | through the whole study, an average of 180 days
  Determination of Number of Participants With Adverse Events

SECONDARY OUTCOMES:
Changing of of virus neutralizing antibody titer | at days 0, 28, 42
  Determination of changing of virus neutralizing antibody titer from baseline scores and at day 28 and 42
Changing of antigen-specific cellular immunity level | at days 0, 10
  Determination of antigen-specific cellular immunity

CONTACTS AND LOCATIONS:
Locations (1):
- ECO-Safety, Saint Petersburg, Russia

IPD SHARING:
Plan to Share IPD: No